CLINICAL TRIAL: NCT01028404
Title: A Trial Investigating the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of NNC 0148-0000-0106 in Healthy Subjects and Subjects With Type 1 and Type 2 Diabetes
Brief Title: A Two Part Trial Investigating NN1952 in Healthy Subjects and Subjects With Type 1 and Type 2 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN1952-3646; U1111-1112-2892 (Other: WHO); 2009-013282-26 (EudraCT Number)
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2; Healthy
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Trial part 1 (Experimental)
  Interventions: Drug: NN1952; Drug: insulin aspart; Drug: placebo
- Trial part 2 (Experimental)
  Interventions: Drug: NN1952; Drug: insulin aspart; Drug: placebo

INTERVENTIONS:
Drug: NN1952 — Subjects will be randomised to receive a single dose of NN1952, at escalating dose levels. Progression to next dose will be based on safety evaluation.
  Arms: Trial part 1
Drug: insulin aspart — As an active comparator, one standard dose will be given s.c. (under the skin) at all dose levels.
  Arms: Trial part 1
Drug: placebo — Subjects will receive a single dose of placebo as a comparator to NN1952, at all dose levels.
  Arms: Trial part 1
Drug: NN1952 — Subjects will be randomised to receive a single dose of NN1952 with or without a meal, on two of four separate study visits. The dose will be selected based on the results of part 1.
  Arms: Trial part 2
Drug: insulin aspart — As an active comparator, one standard dose will be given s.c. (under the skin) at one study visit.
  Arms: Trial part 2
Drug: placebo — Subjects will receive a single dose of placebo as a comparator to NN1952 at one study visit.
  Arms: Trial part 2

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the safety, tolerance, pharmacokinetics (exposure of drug) and pharmacodynamics (effect) of NN1952 as tablets in healthy volunteers and subjects with type 1 and type 2 diabetes.

The trial consists of two parts. In part 1, single escalating doses of NN1952, placebo or insulin aspart will be given to healthy volunteers. In part 2, subjects with type 1 or type 2 diabetes will receive single doses of NN1952 (with/without a meal), insulin aspart and placebo.

ELIGIBILITY:
Inclusion Criteria:

* FOR TRIAL PART 1, THE FOLLOWING APPLIES:
* Gender: male
* Age: 18-55 years
* BMI (body mass index): 18-28 kg/m2
* Study participants considered to be healthy
* FOR TRIAL PART 2, THE FOLLOWING APPLIES:
* Gender: male or female of no childbearing potential
* Age: 18-65 years
* Type 1 diabetes: BMI (body mass index): 18-28 kg/m2
* Type 2 diabetes: BMI (body mass index): 22-35 kg/m2
* Type 1 or type 2 diabetes for at least 12 months
* Type 1 diabetes: Treatment with insulin for at least 12 months
* Type 2 diabetes: Treatment with insulin for at least 3 months

Exclusion Criteria:

* Known or suspected allergy to the trial product or related products
* Presence of illness or infection that may confound the results of the study or pose a risk to the study participant by dosing NN1952, as judged by the Investigator
* Presence of acute gastrointestinal symptoms (for example nausea, vomiting, heartburn or diarrhoea)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2009-11; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events for trial part 1 | from visit 1 to visit 3
Number and severity of adverse events for trial part 2 | from visit 1 to visit 6

SECONDARY OUTCOMES:
Area under the serum insulin concentration-time curve after a single dose | after 12 hours
Area under the glucose infusion rate-time curve after a single dose | after 12 hours

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com